CLINICAL TRIAL: NCT04354038
Title: Host and Bacterial Mechanisms in Recovering FEV1 After Pulmonary Exacerbations in Patients With Cystic Fibrosis
Brief Title: Host and Bacterial Mechanisms During Cystic Fibrosis Pulmonary Exacerbations
Status: Active, not recruiting | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: SAAVED19G0
Record Dates: First submitted 2020-04-13; First posted 2020-04-21 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic fibrosis pulmonary exacerbations (CF PEx) vary greatly in their severity, their pathogens, and their treatment responses. A failure to return to baseline lung function after treatment may be due to persistent infection or chronic inflammation or both. This constant infection and inflammation are believed to be tightly connected, making it difficult to know the exact reason why some patients fail to respond to treatment. The purpose of this study is to evaluate both infection and inflammation during CF PEx to allow for more personalized approaches to improve lung function responses and better CF PEx outcomes. Subjects will be asked to be in the study if they have CF, are 18 years of age or older, and are starting on IV antibiotics due to worsening lung infection. Subjects will stay in the study for up to 5 years, with visits occurring once a year if hospitalized for a CF PEx. Each visit will have blood, sputum, and urine collected and analyzed for changes in expression of certain genes and proteins. These changes may relate to improvements felt by people living with CF and determine what treatments are most helpful.

ELIGIBILITY:
Inclusion Criteria:

* CF patients 18 years or older
* hospitalized for IV treatment of an acute pulmonary exacerbation
* not on investigational drugs
* who can provide written consent and are willing to comply with study procedure

Exclusion Criteria:

• the presence of a condition or abnormality that, in the opinion of the Principal Investigator, would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed by the Colorado Adult CF Center will be eligible. A subject will have a diagnosis of cystic fibrosis, be 18 years or older, and been diagnosed by clinical faculty with a pulmonary exacerbation (PEx) and need to be hospitalized to start on IV antibiotic treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change between FEV1 and Th17/PD-1 expression during the course of treatment for pulmonary exacerbations using flow cytometry | Onset and end of CF pulmonary exacerbations, on average 10 days apart
  There is a Th17 skewing association with a failure to return to baseline FEV1 values post pulmonary exacerbation, as measured using conventional flow cytometry followed by linear mixed effects models.
Change between FEV1 and Th17/PD-1 expression over time using flow cytometry | From initial CF pulmonary exacerbation to subsequent CF pulmonary exacerbation, assessed over a period of 60 months
  There is a Th17 skewing association with a failure to return to baseline FEV1 values post pulmonary exacerbation, as measured using conventional flow cytometry followed by linear mixed effects models.
Change in FEV1 and Th1/Th2/Th17 gene expression during the course of treatment for pulmonary exacerbations using single cell sequencing | Onset and end of CF pulmonary exacerbations, on average 10 days apart
  Gene expression changes, with a particular emphasis on the relationship between changing cell composition (Th1, Th2, and Th17) single cell gene expression and FEV1 recovery, as measured by single cell sequencing of CD4+CD45RO+ memory cells, may be associated with a failure to return to baseline FEV1 during the course of treatment.
Change in FEV1 and Th1/Th2/Th17 gene expression over time using single cell sequencing | From initial CF pulmonary exacerbation to subsequent CF pulmonary exacerbation, assessed over a period of 60 months
  Gene expression changes, with a particular emphasis on the relationship between changing cell composition (Th1, Th2, and Th17) single cell gene expression and FEV1 recovery, as measured by single cell sequencing of CD4+CD45RO+ memory cells, may be associated with a failure to return to baseline FEV1 over time.
Comparison of Th17 vs Th2 TCR repertoires during the course of treatment for pulmonary exacerbations through bulk TCR beta sequencing | Onset and end of CF pulmonary exacerbations, on average 10 days apart
  Examining if an expanded clone within the Th17 lineage translates to greater inflammation and poorer FEV1 response during the course of treatment as measured by bulk TCR beta sequencing.
Comparison of Th17 vs Th2 TCR repertoires over time through bulk TCR beta sequencing | From initial CF pulmonary exacerbation to subsequent CF pulmonary exacerbation, assessed over a period of 60 months
  Examining if an expanded clone within the Th17 lineage translates to greater inflammation and poorer FEV1 response over time as measured by bulk TCR beta sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No